CLINICAL TRIAL: NCT04670393
Title: Impact of the Administration of an Antioxidant Food Supplement Associated With Oral Probiotics on the Ovarian Oxidative Stress Profile and the Intestinal Microbiota Function in the in Vitro Fertilization Cycle of Patients With Polycystic Ovarian Syndrome
Brief Title: Antioxidant Supplement Associated With Oral Probiotics in Patients With PCOS in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fertypharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-FBM+-3
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Infertility, Female; Polycystic Ovary Syndrome
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FertyBiotic Woman Plus (Experimental): Participants received FertyBiotic Woman Plus one sachet a day
  Interventions: Dietary Supplement: FertyBiotic Woman Plus
- Placebo (Placebo Comparator): Participants received 400 mcg of folic acid once a day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: FertyBiotic Woman Plus — 4g Myo-Inositol, 421 mg D-Chiro-Inositol, 400 mcg folic acid, 55 mcg selenium, 15 mcg vitamin D, 1,8 mg melatonin,2x109 Lactobacillus rhamnosus, 2x109 Lactobacillus crispatus and 2x109 Lactobacillus plantarum
  Arms: FertyBiotic Woman Plus
Other: Placebo — 400 mcg folic acid
  Arms: Placebo

SUMMARY:
The aim of the study is to study the effect of an antioxidant food supplement associated with probiotics on the oocyte quality response, oxidative stress and microbiota function in an in vitro fertilization cycle in patients with polycystic ovarian syndrome

DETAILED DESCRIPTION:
After being informed about the study, all patients meeting the inclusion/exclusion criteria and giving written informed consent will be randomized in a double-blind manner in a ratio 1:1 to receive the antioxidant supplementation associated with probiotics (Myo-Inositol, D-Chiro-Inositol, folic acid, selenium, vitamin D, Melatonin, Lactobacillus rhamnosus, Lactobacillus cripatus and Lactobacillus plantarum) or placebo (folic acid) once daily.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-38 years old
* Diagnosis of PCOS according to compliance with the Rotterdam criteria
* BMI >= 25

Exclusion Criteria:

* Hormonal contraceptive, insulin sensitizers such as metformin, inositols, antioxidants, vitamin supplements except folic acid, GnRH analogs, steroidal drugs or others with anti-inflammatory properties, antibiotics, probiotics, laxatives use in the 3 months prior to recruitment
* Tobacco consumption in last 12 months
* Endometriosis, hydrosalpinx not surgically treated, acute or chronic inflammatory diseases, systemic immune diseases, other endocrine diseases or dysfunctions except for PCOS and subclinical hypothyroidism treated with low doses of levothyroxine (eg congenital adrenal hyperplasia, Cushing's syndrome, androgen-secreting tumors, Diabetes Millitus, hyperprolactinemia, hyperglycemia), active neoplastic disease or without evidence of complete remission for at least 5 years,
* Active participation in an active weight reduction program or hypocaloric diet during the study period. No change in habits will be taught during the study period
* Hypersensitivity to any of the components in the Fertybiotic Mujer Plus® formulation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Number of MII oocytes | 3 months in follicular puncture visit

SECONDARY OUTCOMES:
Glucose | Baseline and about 2,5 months when the cycle treatment starts
  Blood glucose
Insulin | Baseline and about 2,5 months when the cycle treatment starts
  Blood glucose
FSH | Baseline and about 2,5 months when the cycle treatment starts
  Follicle Stimulating Hormone in blood
LH | Baseline and about 2,5 months when the cycle treatment starts
  Luteinizing Homone in blood
Testosterone | Baseline and about 2,5 months when the cycle treatment starts
  blood testosterone
Androstendione | Baseline and about 2,5 months when the cycle treatment starts
  blood androstendione
MDA | Baseline (plasma) and 3 months in follicular puncture visit (plasma and follicular puncture)
  Malondialdehyde (MDA) in plasma and follicular liquid
TAC | Baseline (plasma) and 3 months in follicular puncture visit (plasma and follicular puncture)
  Total Antioxidant Capacity (TAC) in plasma and follicular liquid
8-OH-desoxiguanosin | 3 months in follicular puncture visit
  8-OH-desoxiguanosin in granulose cells
Glutation | 3 months in follicular puncture visit
  Glutation in granulose cells
Sirtuin | 3 months in follicular puncture visit
  Sirtuin in granulose cells
Zonulin | Baseline and about 2,5 months when the cycle treatment starts
  Determination of zonulin in plasma
SCFA | Baseline and about 2,5 months when the cycle treatment starts
  Determination of Short-Chain Fatty Acids (SCFA) in feces
Gonadotropin UI | 3 months in follicular puncture visit
Follicles | 3 months in follicular puncture visit
  Number of follicles >= 11 mm in trigger day
Stimulation days | 3 months in follicular puncture visit
Oocytes | 3 months in follicular puncture visit
  Number of oocytes obtained, transferred and frozen
Pregnancy rate | Through study completion, an average of 1 year
Live birth rate | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No